CLINICAL TRIAL: NCT00013117
Title: Computer-Assisted Access to Specialist Expertise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: VCR 99-008
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Telephone specialist consultation

INTERVENTIONS:
Behavioral: Telephone specialist consultation

SUMMARY:
The goal of this research was to determine if providing specialist input to primary care providers (PCPs) by means of informal consultation could improve the process and outcomes of care for diabetes. Several studies support the role for specialists and their specific knowledge and expertise in a variety of disorders including diabetes. A variety of methods have been designed to optimize the use of specialty expertise including practice guidelines and disease management approaches as well as the consultation/referral process. The referral-consultation process is an important mechanism for obtaining clinically useful information. At one end of the spectrum of this process, informal consultation involves discussion about a patient with a colleague without the consultant seeing the patient; at the other end of the spectrum, care of the patient is transferred to another physician and the process is formalized. Because much specialist expertise resides in the specialists themselves, the expansion of primary care sites to include community-based outpatient clinics has implications for access to the specialists located elsewhere. This study was designed to evaluate a computer-assisted voice mail system which is relatively inexpensive and more convenient than video-telemedicine systems, making it more practical and more easily exportable. Diabetes care delivery was chosen as the model in which to assess informal consultation based on its frequency among veterans, management challenges, and the emphasis on improvement in diabetes care in VA. A secondary goal of the project was to better characterize the consultation process.

DETAILED DESCRIPTION:
Background:

The goal of this research was to determine if providing specialist input to primary care providers (PCPs) by means of informal consultation could improve the process and outcomes of care for diabetes. Several studies support the role for specialists and their specific knowledge and expertise in a variety of disorders including diabetes. A variety of methods have been designed to optimize the use of specialty expertise including practice guidelines and disease management approaches as well as the consultation/referral process. The referral-consultation process is an important mechanism for obtaining clinically useful information. At one end of the spectrum of this process, informal consultation involves discussion about a patient with a colleague without the consultant seeing the patient; at the other end of the spectrum, care of the patient is transferred to another physician and the process is formalized. Because much specialist expertise resides in the specialists themselves, the expansion of primary care sites to include community-based outpatient clinics has implications for access to the specialists located elsewhere. This study was designed to evaluate a computer-assisted voice mail system which is relatively inexpensive and more convenient than video-telemedicine systems, making it more practical and more easily exportable. Diabetes care delivery was chosen as the model in which to assess informal consultation based on its frequency among veterans, management challenges, and the emphasis on improvement in diabetes care in VA. A secondary goal of the project was to better characterize the consultation process.

Objectives:

Patients with diabetes mellitus are complex and may benefit from the input of multiple specialists and PCPs must determine the need for and coordinate the input from those multiple specialists. With that in mind, the three objectives of the study are: 1) To assess the impact of computer-assisted access to specialist expertise (CASE) on process of care for patients with diabetes mellitus; 2) To assess the impact of CASE on outcomes of care at the patient level (clinical outcomes and satisfaction), provider level (satisfaction) and the system level (health services utilization and costs); and 3) To characterize the consultation-referral process in community-based outpatient clinics (CBOCs).

Methods:

Randomized controlled trial with access to the CASE system constituting the intervention and a descriptive study of the consultation process. The major outcome variables will be the consultation type, adherence to diabetes practice guidelines, clinical outcome of diabetes care (glycemic control), patient and provider satisfaction.

Status:

Project work has been completed. The final report has been submitted.

ELIGIBILITY:
Inclusion Criteria:

Primary Care Providers in VA community-based outpatient clinics; patients receiving primary care in VA community-based outpatient clinics.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Aron, MD MS, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States